CLINICAL TRIAL: NCT02826551
Title: Pain Outcomes After Anterior Cruciate Ligament Reconstruction With Posterior Capsular Marcaine Injection: A Prospective Randomized Trial
Brief Title: Pain Outcomes After Anterior Cruciate Ligament Reconstruction With Posterior Capsular Marcaine Injection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough data.
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Michael Banffy, Attending - PI, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro41651
Record Dates: First submitted 2016-05-24; First posted 2016-07-11 (Estimated); Results first posted 2017-12-14 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Anesthesia
MeSH Terms: interventions — Bupivacaine; Ice; oxycodone-acetaminophen; Crutches

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Injection (Placebo Comparator): These patients will receive standard of care when undergoing anterior cruciate ligament reconstruction and will NOT be receiving a posterior capsular knee injection of Marcaine 0.5%.
  They will be monitored for pain control and pill intake while in the PACU and the first four days post-operatively the same as the patients in the INJECTION Arm of the study.
  Interventions: Other: Ice; Drug: Percocet; Device: Knee Brace and Crutches
- Injection (Experimental): These patients will receive standard of care when undergoing anterior cruciate ligament reconstruction but will additionally be receiving a one-time posterior capsular knee injection of Marcaine 0.5% (20cc) during the surgery.
  They will be monitored for pain control and pill intake while in the PACU and the first four days post-operatively the same as the patients in the NO injection Arm of the study.
  Interventions: Drug: Marcaine; Other: Ice; Drug: Percocet; Device: Knee Brace and Crutches

INTERVENTIONS:
Drug: Marcaine — Pain control medication to theoretically reduce the amount of posterior knee pain that is common after ACL surgery by placing the injection into the posterior capsule of the knee during surgery. This is very easy and safe to accomplish as the surgeon will have direct visualization of the posterior capsule during the surgery.
  Arms: Injection
Other: Ice
Drug: Percocet
Device: Knee Brace and Crutches

SUMMARY:
Post-operative pain control following elective anterior cruciate ligament reconstruction continues to be a hurdle for orthopaedic surgeons. This obstacle becomes particularly problematic during the first 36 hours after the operation, when the patient is experiencing pain at its peak intensity. Good control of pain leads to better patient comfort, confidence to place weight on the operative limb and improved ability to perform critical exercises in this period to improve joint range of motion.

A variety of anesthetic techniques have been employed to reduce pain including: cryotherapy, systemic analgesic and anti-inflammatory drugs, intrathecal, regional blockade of peripheral nerves and frequently intra-articular injections. Each technique has been studied at length with mixed but overall favorable results. However, in the authors' experience, after femoral nerve blockade, patients continue to complain of posterior knee pain in the Post-Anesthesia Care Unit (PACU) and peri-operative period. Intra-articular injections comprised of morphine and other Na-channel blocker analgesics may curb some of this pain by bathing the posterior capsule in anesthetic. However, there is still a large concern amongst orthopaedic surgeons about the potential harm these agents may have on the knee's healthy articular cartilage surfaces. The long term effects, including chondrolysis have been documented in the shoulder and while in the short term this effect is diminished there is still hesitation among surgeons to use this form of pain blockade.

This has led the investigators to adapt a technique of isolated posterior capsular injections after total knee replacements from the joint arthroplasty literature, which has shown favorable results with low complication risk. The investigators plan to study the effectiveness of this technique during ACL reconstruction in an attempt to curb the amount of posterior knee pain and decrease the overall narcotic use postoperatively while limiting the exposure of the native cartilage to harmful agents.

DETAILED DESCRIPTION:
A prospective series of consecutive patients undergoing primary ACLR will be recruited from a preoperative log of patients seeing one of two sports medicine fellowship trained surgeons within the investigators group. Patients undergoing primary unilateral anterior cruciate ligament reconstruction (ACLR) either with bone-patellar bone autograft or Achilles tendon allograft will be included by surgeons using similar techniques and fixation options.

After consenting to participate, subjects will be randomized into one of two groups. Using a random number generator, 60 consecutively enrolled patients will be placed in their appropriate study arm. (Odd numbers = Control Group) (Even numbers = Experimental Group). Only the patient will be blinded to which arm of the study they belong.

Group 1(Control) patients will undergo routine arthroscopically assisted ACLR surgery with a standardized postoperative protocol. Group 2 (Experimental) patients will undergo the same procedure with the same postoperative protocols as Group 1, with the addition of the posterior capsular injection of 20 cc of Marcaine 0.5%. There are no placebo treatments being offered and the surgeons and operating room staff are not blinded to the subjects group. Injecting marcaine in this study will be performed in accordance with its standard use according to the FDA labeling/guidelines. The physicians will use their discretion as to the appropriate location for the injection into the posterior capsule of the knee which should bring no additional risks than expected for a knee injection.

At the conclusion of the case, each patient will receive a dry sterile dressing, followed by a compression wrap and a hinged knee brace locked in extension. No drains, pain pumps or nerve stimulators will be used. The nurses in the recovery room who will be administering the VAS assessment and recording time and frequency of pain medication dosing will be blinded to the patients' Group number. The nurses will provide pain medications and the visual analog assessment for their duties in the post-op anesthesia unit, and are not administering drugs or procedures specifically for research purposes.

Post-operative Care All patients will be discharged home from the surgery center on the same day (within 2-3 hours) postoperatively. Patients will be made weight bearing as tolerated with crutches and a brace.

While in the PACU, at time points 15min and 1 hour, a standardized and previously validated visual analog scale (VAS) for pain assessment will be delivered to the patient by the recovery room nurse.

Patients after discharge will then be asked to rate their most severe pain each morning and night for 4 consecutive postoperative days using this VAS pain scale. A standardized pain medication regimen will be given including: one or two tabs of Percocet 7.5/325mg to be taken every 4 to 6 hours as needed. A log of the time and amount of medication taken each POD will be kept and recorded by the patients. Patients will also be instructed to use cryotherapy for 20 min intervals 3 times per day. Patients will also begin on POD 0 the use of continuous passive motion machines starting at a comfortable range of motion and progressing 5 degrees/day as tolerated. Patients will return for their first post-operative visit between 7-10 days where diaries will be collected and the patient clinically assessed.

Patient's will also be seen at their three month post-operative visit and be clinically assessed for the presence of chondrolysis (a frequently measured outcome during knee pain medication injection studies).

Statistical Analysis Based on previous studies, the Mann-Whitney U test will check differences between numeric variables. Nonparametric Kruskal-Wallis tests can compare the analgesia level in the two groups and if possible ANOVA test can compare the analgesia duration. Chi-square tests will be utilized for any potential complications which will also be recorded.

Power Analysis Prelim Power Analysis per STATS department @ Cedars: sample sizes of 26 for each group (N1=N2=26) = Total 52 patients to achieve 80% power to reject the null hypothesis of equal means when the population mean difference is 2 with a standard deviation for both groups of 2.5 and with a significance level (alpha) of 0.050 using a two-sided two-sample equal-variance t-test. A total of 60 patients will be enrolled to ensure the investigators achieve adequate power for the study.

Despite the addition of selective regional blockade by the anesthesia team including femoral and saphenous nerve blocks, a portion of patients are still experiencing post-operative knee pain within the first few hours to days after the procedure. Pain may be a result of the femoral tunnel drilling which theoretically may be relieved by a posterior capsular injection. Eliminating this painful period will improve the patient's subjective experience undergoing surgery, and may also allow for earlier range of motion and participation in rehabilitation strengthening exercises performed by the patient in the peri-operative period.

ELIGIBILITY:
Inclusion Criteria:

* Adult individuals (ages 18-60), both sexes, submitted to elective ACL reconstructions with or without partial menisectomies of the medial or lateral meniscus

Exclusion Criteria:

* Multiligamentous injury or revision surgery
* Known narcotic/substance abuse or regular opiate use
* Known allergy to any medication or anesthetic being used in this study
* Patients with pre-existing diabetic or femoral neropathy
* INTRAOPERATIVELY- if chrondral microfractures, inside-out or outside-in meniscal repairs were performed (***Since these additional surgeries within the joint may increase the perceived level of pain post-op***)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2017-05-10 (Actual)

REFERENCES:
- [Background] Guild GN 3rd, Galindo RP, Marino J, Cushner FD, Scuderi GR. Periarticular regional analgesia in total knee arthroplasty: a review of the neuroanatomy and injection technique. Orthop Clin North Am. 2015 Jan;46(1):1-8. doi: 10.1016/j.ocl.2014.09.016. PMID 25435030

RESULTS

PARTICIPANT FLOW:
Groups:
- No Injection: These patients will receive standard of care when undergoing anterior cruciate ligament reconstruction and will NOT be receiving a posterior capsular knee injection of Marcaine 0.5%.
  They will be monitored for pain control and pill intake while in the PACU and the first four days post-operatively the same as the patients in the INJECTION Arm of the study.
  Ice
  Percocet
  Knee Brace and Crutches
- Injection: These patients will receive standard of care when undergoing anterior cruciate ligament reconstruction but will additionally be receiving a one-time posterior capsular knee injection of Marcaine 0.5% (20cc) during the surgery.
  They will be monitored for pain control and pill intake while in the PACU and the first four days post-operatively the same as the patients in the NO injection Arm of the study.
  Marcaine: Pain control medication to theoretically reduce the amount of posterior knee pain that is common after ACL surgery by placing the injection into the posterior capsule of the knee during surgery. This is very easy and safe to accomplish as the surgeon will have direct visualization of the posterior capsule during the surgery.
  Ice
  Percocet
  Knee Brace and Crutches
Period: Overall Study
Arm/Group | No Injection | Injection
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Number of Participants Consented
Groups:
- Total: Total of all reporting groups
Arm/Group | No Injection | Injection | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 23
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 6 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 12 | 23
Subjects Injected or Not Injected [Number; unit: participants] | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: VAS Scores
Description: VAS Scales recorded in AM and PM
Time Frame: Day 0-4 post-operatively
Population: data were not collected.
Arm/Group | No Injection | Injection
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Pain Pill Count
Description: Patients will log the number of pills they take the first four days after surgery.
Time Frame: Day 0-4 post-operatively
Population: data was not collected.
Arm/Group | No Injection | Injection
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year.
Arm/Group | No Injection | Injection
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 0/11 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2015-07-01): https://cdn.clinicaltrials.gov/large-docs/51/NCT02826551/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-26): https://cdn.clinicaltrials.gov/large-docs/51/NCT02826551/SAP_001.pdf